CLINICAL TRIAL: NCT03808389
Title: A Double-blind, Placebo-controlled, Randomized Clinical Trial Investigating Fecal Microbiota Transplantation for Parkinson's Disease and Its Effect on Symptoms and Disease Progression
Brief Title: Fecal Microbiota Transplantation for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other); the Flanders Institute for Biotechnology (Unknown); Research Foundation Flanders (Other); Vlaamse Parkinson Liga (Unknown); Parkili (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGent2018/0623
Record Dates: First submitted 2018-06-22; First posted 2019-01-17 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Fecal microbiota transplantation; Microbiome; Gut-brain axis
MeSH Terms: conditions — Parkinson Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: 40 patients with Parkinson's disease (Hoehn & Yahr score 2-3) will be randomly allocated (20 vs. 20) to either fecal microbiota transplantation with donor stool or autologous fecal microbiota transplantation (= own stool).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group: Donor FMT (Experimental): Fecal microbiota transplantation using fecal matter from a healthy donor selected through strict inclusion criteria assessing the presence of any infectious diseases.
  Interventions: Other: Donor FMT
- Control group: Autologous FMT (Sham Comparator): Fecal microbiota transplantation using the patient's own fecal matter.
  Interventions: Other: Autologous FMT

INTERVENTIONS:
Other: Donor FMT — Fecal microbiota transplantation through nasojejunal administration. Fecal matter will be collected prior to the start of the study from healthy donors and will be frozen at -80°C after thorough screening for infectious diseases. At the time of transplantation, samples will be thawed and administrated to the patients in the treatment group.
  Other Names: FMT with donor stool
  Arms: Treatment group: Donor FMT
Other: Autologous FMT — Fecal microbiota transplantation through nasojejunal administration. Fecal matter will be collected prior to the start of the study from each patient and will be frozen at -80°C after thorough screening for infectious diseases. At the time of transplantation, samples will be thawed and administrated to the patients in the control group.
  Other Names: FMT with own stool
  Arms: Control group: Autologous FMT

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder and due to the lack of early diagnosis and effective therapy, represents a large burden for our society and healthcare system. The last years, it became increasingly apparent that non-motor symptoms, including gastrointestinal dysfunction, precede the onset of the typical PD motor symptoms by several years. Moreover, emerging evidence suggests that PD, and more specifically the aggregation of alpha-synuclein, starts in the gut before spreading to the brain. Additionally, recent microbiome studies consistently showed microbiota differences between PD patients and healthy controls.

The ultimate goal of this project is to address the impact of gut dysbiosis and the restoration of gut homeostasis by fecal microbiota transplantation (FMT) on the development and progression of PD. We will identify PD-specific changes in microbiota composition and gut inflammation and determine the effect of a 'microbiome-reset' approach through FMT in PD patients on the identified changes and more importantly on disease symptoms and progression.

DETAILED DESCRIPTION:
In this study the effects of fecal microbiota transplantation (FMT) on patients with Parkinson's disease will be investigated in a double-blind, placebo-controlled randomized clinical trial.

At time of FMT, forty patients will be randomized in a double-blinded fashion to the treatment arm (healthy donor stool) or placebo arm (own stool). Transplantation will be performed through nasojejunal administration.

Donors for this study will be recruited from a healthy donor pool who will donate stool after clearance of a strict inclusion protocol which will assess the presence of any infectious diseases. Donor stool will be frozen and stored until day of FMT.

Participants will be screened for relevant inclusion and exclusion criteria and will have to sign an informed consent before admission to the study.

Prior and on a regular basis following the FMT participants will be evaluated through neurological clinical examination and standardized clinical scoring scales including MDS-UPDRS, PDQ-39, NMSS and MoCA. Stool samples will be taken regularly and stored at -80°C for microbiome analysis. Blood will be collected for determining relevant markers. All participants will also undergo sampling for oral and nasal microbiome. Follow-up will continue for a total duration of one year.

Prior to FMT, all participants will undergo a colonoscopy to exclude contra-indications for FMT and to collect mucosa-adherent microbial samples and gastrointestinal tissue biopts. This colonoscopy will be repeated once, one year following the FMT.

The primary endpoint in this study will be a change in clinical status measured through the MDS-UPDRS. Additionally, motor and non-motor symptoms will be correlated with serum markers of inflammation and gut and central nervous system barrier function, microbiota changes and gastrointestinal biopsy analysis of inflammation.

ELIGIBILITY:
Inclusion Criteria for patients:

* Signed informed consent.
* Clinical PD diagnosis (MDS criteria)
* Hoehn & Yahr score of 2-3 in OFF
* Age of motor symptoms onset > 50 years

Exclusion Criteria for patients:

* First degree relative or more than one relative with PD
* Diagnosis of dementia or MMSE < 25
* Diagnosis of major depression or psychosis (DSM-V criteria)
* Any of the following within the previous 2 months: hospital admission, narcosis or sedation, abdominal trauma
* Primary disease of gastrointestinal tract (exception: chronic gastritis)
* Previous abdominal or anorectal surgery (causing structural abnormalities of the intestines)
* Any of the following within the previous 2 months: gastrointestinal or respiratory tract infection, food intoxication
* The use of probiotics or antibiotics within three months prior to FMT
* Contra-indications for colonoscopy
* Other immune disorder or clinical immunosuppression
* Drug abuse
* Malignancy
* Any severe comorbidity that might interfere with the study course as determined by the treating physician
* Pregnancy or inadequate anti conception for the duration of the trial

Inclusion criteria for donors

* age 18 - 75 years
* signed informed consent
* normal screening protocol, including screening for infectious diseases, according to the recommendations of the Superior Health Council of Belgium concerning the safety and quality of fecal transplantation in humans

Exclusion criteria for donors

* presence of gastrointestinal symptoms
* gastro-intestinal or other important comorbidity
* obesity or metabolic syndrome
* history of malignancy both gastrointestinal or systemic
* presence of known colon polyps
* recent placing of piercings/tattoos
* sexual risk behaviour
* antimicrobial therapy 3 months prior to donation
* living in the same household as a Parkinson's disease patient

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Changes in clinical symptoms as scored on the MDS-UPDRS (Movement Disorder Society - Unified Parkinson's Disease Rating Scale) | 3 months, 6 months, 12 months
  The MDS-UPDRS (Movement Disorder Society - Unified Parkinson's Disease Rating Scale) has four parts: Part I (non-motor experiences of daily living; 13 items), Part II (motor experiences of daily living; 13 items), Part III (motor examination; 33 scores based on 18 items, several with right, left or other body distribution scores) and Part IV (motor complications; 6 items). Each item has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Part III will be clinically scored in an OFF-medication state. Subscales are analyzed separately.
  References:
  1. Goetz, C. et al. Movement Disord 22, 41-47 (2007).
  2. Goetz, C. et al. Movement Disord 23, 2129-2170 (2008).

SECONDARY OUTCOMES:
Changes in non-motors symptoms as scored on the Non-motor symptoms scale for Parkinson's disease (NMSS) | 3 months, 6 months, 12 months
  Non-motor symptoms scale for Parkinson's disease (NMSS). Non-motor symptoms are assessed over the last month. Each symptom is scored with respect to:
  Severity: 0 = None; 1 = Mild: symptoms present but causes little distress or disturbance to patient; 2 = Moderate: some distress or disturbance to patient; 3 = Severe: major source of distress or disturbance to patient.
  Frequency: 1 = Rarely (<1/wk); 2 = Often (1/wk); 3 = Frequent (several times per week); 4 = Very Frequent (daily or all the time).
  NMSS contains nine dimensions: cardiovascular (2 items), sleep/fatigue (4 items), mood/cognition (6 items), perceptual problems (3 items), attention/memory (3 items), gastrointestinal (3 items), urinary (3 items), sexual function (2 items), and miscellaneous (4 items).
  Subscores are calculated through multiplication of frequency x severity. Total score is calculated by adding all subscores, range 0-360.
  Reference: Chaudhuri, K. R. et al. Mov. Disord. 22, 1901-11 (2007).
Changes in quality of life as scored on the Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 3 months, 6 months, 12 months
  Parkinson's Disease Quality of Life Questionnaire. All 39 questions are coded in the same way: 0 = Never; 1 = Occasionally; 2 = Sometimes; 3 = Often; 4 = Always (or cannot do at all, if applicable).
  The different dimensions are mobility (10 items), activities of daily living (6 items), emotional well being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items).
  Each dimension is calculated as a scale from 0 to 100 (0 = no problem at all; 100 = maximum level of problem). Formula for scoring each dimension = (sum of scores of each question in dimension)/ (4 x number of questions in dimension) x 100.
  The Single Index score: PDQ-SI= summing the eight dimensions and then dividing by eight.
  Reference: Jenkinson, C., Fitzpatrick, R., Peto, V., Greenhall, R. & Hyman, N. Age Ageing 26, 353-7 (1997).
Changes in cognition as scored on the Montreal Cognitive Assessment (MoCA) | 3 months, 6 months, 12 months
  The Montreal Cognitive Assessment (MoCA) assesses several cognitive domains: short-term memory, visuospatial abilities, executive functions, attention, concentration, working memory, language, orientation to time and place. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.
  Reference: Nasreddine, Z. et al. J Am Geriatr Soc 53, 695-699 (2005).
Number of participants with a change in required anti-PD symptomatic or levodopa therapy | 3 months, 6 months, 12 months
Changes in gastrointestinal symptoms as assessed by the Rome IV questionnaire | 3 months, 6 months, 12 months
  The Rome IV criteria for functional constipation and irritable bowel syndrome are assessed to evaluate potential change in gastrointestinal symptoms following the fecal microbiota transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Santens, MD, PhD, Principal Investigator — Ghent University, Ghent University Hospital
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruggeman A, Vandendriessche C, Hamerlinck H, De Looze D, Tate DJ, Vuylsteke M, De Commer L, Devolder L, Raes J, Verhasselt B, Laukens D, Vandenbroucke RE, Santens P. Safety and efficacy of faecal microbiota transplantation in patients with mild to moderate Parkinson's disease (GUT-PARFECT): a double-blind, placebo-controlled, randomised, phase 2 trial. EClinicalMedicine. 2024 Mar 27;71:102563. doi: 10.1016/j.eclinm.2024.102563. eCollection 2024 May. PMID 38686220